CLINICAL TRIAL: NCT03302104
Title: Diet Quality Indices and Leukocyte Telomere Length Among Healthy US Adults: Data From the National Health and Nutrition Examination Surveys (NHANES) 1999-2002
Brief Title: Diet Quality and LTL in NHANES
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: R01AG033592-01A1 (NIH)
Record Dates: First submitted 2017-09-22; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Telomere Length, Mean Leukocyte; Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our study, we used data from 4,758 healthy adults from the 1999-2002 National Health and Nutrition Examination Surveys to examine the associations between evidence-based diet quality indices and leukocyte telomere length. Our study assessed the four most widely recognized and commonly used diet quality indices in nutritional epidemiology: the USDA-developed Healthy Eating Index-2010, the Alternate Healthy Eating Index-2010, the Mediterranean Diet Score, and the DASH diet score. Analyses were adjusted for sociodemographic and health variables known to influence dietary intake and cellular aging.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20 to 65 years
* No prior diagnosis of major chronic disease (coronary heart disease, angina, myocardial infarction, stroke, diabetes, congestive heart failure, and cancer)

Exclusion Criteria:

* Prior diagnosis of major chronic disease (coronary heart disease, angina, myocardial infarction, stroke, diabetes, congestive heart failure, and cancer)
* Younger than age 20 or older than age 65

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population was comprised of 4,758 healthy adults, aged 20 to 65 years, who had complete dietary and leukocyte telomere length (LTL) data measured in 1999-2002 National Health and Nutrition Examination Surveys (NHANES), without a prior diagnosis of major chronic disease (coronary heart disease, angina, myocardial infarction, stroke, diabetes, congestive heart failure, and cancer).
Sampling Method: Probability Sample
Enrollment: 4758 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2002-12-31 (Actual); Study Completion 2002-12-31 (Actual)

PRIMARY OUTCOMES:
Leukocyte telomere length | 1999-2002